CLINICAL TRIAL: NCT04937283
Title: Comparison of Segmentectomy Versus Lobectomy for Lung Adenocarcinoma ≤ 2cm With Micropapillary and Solid Subtype Negative by Intraoperative Frozen Sections: A Prospective and Multi-center Randomized Controlled Trial Study
Brief Title: Segmentectomy Versus Lobectomy for Lung Adenocarcinoma ≤ 2cm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Deping Zhao, Director of Thoracic Surgery, Shanghai Pulmonary Hospital, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAR001
Record Dates: First submitted 2021-04-24; First posted 2021-06-24 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Lung Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Mastectomy, Segmental

STUDY DESIGN:
Intervention Model Description: segmentectomy group versus lobectomy group
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Segmentectomy with systemic lymph node dissection (Experimental): Segmentectomy with hilar and mediastinal lymph node dissection is performed. If the tumor located at inter-segment plane and without sufficient resection margin distance, a combined segmentectomy will be performed after a comprehensive evaluation. As with lobectomy, systemic or selective lymph node dissection is mandatory, and nodal sampling is not allowed. At least three stations of mediastinal lymph node from 2R, 4R, 7, 8, 9 for the right side and 5, 6, 7, 8, 9 for the left side, respectively. The distance from the dissection margin to the tumor edge must be evaluated in the same manner as with lobectomy. When lymph node metastasis is present or resection margin is not cancer-free, the surgical procedure must be converted to a lobectomy.
  Interventions: Procedure: Segmentectomy with systemic lymph node dissection
- Lobectomy with systemic lymph node dissection (Active Comparator): lobectomy with hilar and mediastinal lymph node dissection is performed. Systemic or selective lymph node dissection is mandatory, and nodal sampling is not allowed. At least three stations of mediastinal lymph node from 2R, 4R, 7, 8, 9 for the right side and 5, 6, 7, 8, 9 for the left side, respectively.
  The distance from the dissection margin to the tumor edge must be evaluated intraoperatively. If the distance is either less than the maximum tumor diameter or ,20 mm, the absence of cancer cells in the resection margin must be histologically or cytologically confirmed before finishing surgery.
  Interventions: Procedure: Lobectomy with hilar and mediastinal lymph node dissection

INTERVENTIONS:
Procedure: Segmentectomy with systemic lymph node dissection — Segmentectomy with hilar and mediastinal lymph node dissection is performed. If the tumor located at inter-segment plane and without sufficient resection margin distance, a combined segmentectomy will be performed. Systemic or selective lymph node dissection is mandatory, and nodal sampling is not allowed. At least three stations of mediastinal lymph node from 2R, 4R, 7, 8, 9 for the right side and 5, 6, 7, 8, 9 for the left side, respectively. The distance from the dissection margin to the tumor edge must be evaluated intra-operatively. If the distance is either less than the maximum tumor diameter or 20 mm, the absence of cancer cells in the resection margin must be histologically or cytologically confirmed before finishing surgery.
  Arms: Segmentectomy with systemic lymph node dissection
Procedure: Lobectomy with hilar and mediastinal lymph node dissection — Lobectomy with hilar and mediastinal lymph node dissection is performed. Segmentectomy with hilar and mediastinal lymph node dissection is performed. Systemic or selective lymph node dissection is mandatory, and nodal sampling is not allowed. At least three stations of mediastinal lymph node from 2R, 4R, 7, 8, 9 for the right side and 5, 6, 7, 8, 9 for the left side, respectively. The distance from the dissection margin to the tumor edge must be evaluated intra-operatively. If the distance is either less than the maximum tumor diameter or 20 mm, the absence of cancer cells in the resection margin must be histologically or cytologically confirmed before finishing surgery.
  Arms: Lobectomy with systemic lymph node dissection

SUMMARY:
This study aims to evaluate the non-inferiority in recurrence-free survival and overall survival of segmentectomy compared with lobectomy in patients with lung adenocarcinoma ≤ 2 cm with micropapillary and solid subtype negative by intraoperative frozen sections.

DETAILED DESCRIPTION:
At present, the technology of intraoperative frozen section has gradually matured, which can diagnose the benign and malignant tumors and guide the resection strategy for peripheral small-sized lung adenocarcinoma. Travis et al. reported high specificity of intraoperative frozen section in the identification of micropapillary components, confirming that intraoperative frozen section may guide the selection of surgical procedures. However, there is still little evidence weather segmentectomy is appropriate for invasive adenocarcinoma without micropapillary patterns. This prospective and multi-center study was aimed to evaluate the non-inferiority in recurrence free survival and overall survival of segmentectomy compared with lobectomy in patients with lung adenocarcinoma (≤ 2 cm) not including micropapillary components.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 20-79 years old, both male or female;
* Tumor size <= 2cm on preoperative CT scan;
* Peripheral solitary nodule or the associated lesion is MIA or less invasive lesion;
* Preoperative CT indicated that the nodules were non-pure glass nodules (consolidation to tumor ratio >= 0.25);
* Intraoperative frozen section confirmed invasive lung adenocarcinoma with micropapillary and solid subtype negative (<= 5%);
* Intraoperative frozen section indicated the resection margins was free of tumor cells;
* Lung function could withstand both lung segmentectomy and lobectomy (FEV1 > 1.5L or FEV1% >= 60%);
* Eastern Cooperative Oncology Group, 0 to 2;
* Volunteer to participate the trial and sign the informed consent, able to comply with the follow-up plan and other program requirements.

Exclusion Criteria:

* Radiological pure ground glass nodules (consolidation to tumor ratio < 0.25);
* The nodule is close to the lung hilus and is unable to perform segmentectomy;
* Intraoperative frozen section confirmed with micropapillary and solid subtype positive (> 5%);
* Intraoperative frozen section confirmed adenocarcinoma in situ and minimally invasive adenocarcinoma;
* Preoperative imaging examination or EBUS indicated lymph node positive metastasis;
* Preoperative imaging examination revealed distant metastasis;
* Patients with severe damage to heart, liver and kidney function (grade 3 ~ 4, ALT and/or AST over 3 times the normal upper limit, Cr over the normal upper limit);
* Patients with other malignant tumors;
* Pregnant, planned pregnancy and lactating female patients (urine HCG>2500IU/L is diagnosed as early pregnancy);
* Prior chemotherapy, radiation therapy or any other therapies were performed; 12 participated in other tumors within three months of relevant clinical subjects;
* Those who have participated in other tumor-related clinical trials within three months;
* Those are not suitable for participating in trials according to investigator's assessment.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
recurrence-free survival rate | 5 year
  Recurrence-free survival (RFS) was defined as the time from surgery until recurrence or death from any cause

SECONDARY OUTCOMES:
overall survival | 5 year
  Overall survival (OS) was defined as the time from surgery until death from any cause
Post-operative respiratory function | 6 months
  The post-operative respiratory function will be evaluated by FEV1% and FVC.
Operation time | 24 hours
  The surgery time in both groups.
Blood loss | 24 hours
  Intraoperative blood loss in total.
Incidence of operative complications | 1 month
  Any intraoperative complications related to the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Chen, MD, PhD, Principal Investigator — Shanghai Pulmonary Hospital, School of Medicine, Tongji University
Locations (14):
- China (14):
  - Anhui Chest Hospital, Hefei, Anhui
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Nanyang Central Hospital, Nanyang, Henan
  - The Sixth People's Hospital of Nantong, Nantong, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Yancheng First People's Hospital, Yancheng, Jiangsu
  - Shandong Public Health Clinical Center, Jinan, Shandong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Huadong Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Ningbo No.2 Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No